CLINICAL TRIAL: NCT01020435
Title: Upper Cervical Manipulation for Patients With Stage 1 Hypertension
Brief Title: Chiropractic for Hypertension in Patients
Acronym: CHiP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHiP; NCT01230372 (obsolete NCT alias)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Manipulation, Spinal; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal Manipulation High Velocity (Active Comparator): This non-rotary upper cervical procedure uses an impulse thrust with a controlled depth (high velocity). The participant's head is supported by a specially designed cushion and the doctor usually approaches the participant from in front of his or her head to contact soft tissue over the atlas transverse process, posterior to the lateral mass or occasionally on the C2 lamina or spinous process, with the pisiform process of one hand. The thrust is delivered by a contraction of the triceps muscles of both arms, which straightens the arms and applies the thrust to the participant.
  Interventions: Other: Spinal Manipulation
- Sham Spinal Manipulation (Placebo Comparator): The sham assessment procedures will be similar to the active group. It has been developed and validated by Vernon et al.
  Interventions: Other: Sham Spinal Manipulation

INTERVENTIONS:
Other: Spinal Manipulation — The procedure in its broadest definition describes the application of a load (force or displacement) to specific body tissues (usually vertebral joints) with therapeutic intent. The mechanical characteristics of SM can vary in terms of its duration and amplitude, (hence, the rate at which it is applied), as well as its anatomical location, choice of levers, direction of force application, and the vehicle used to apply the force (manually or mechanically assisted).
  Arms: Spinal Manipulation High Velocity
Other: Sham Spinal Manipulation — The sham assessment procedures will be the same as those in the high velocity treatment group. The sham intervention is identical to this treatment protocol except for the placement of the treating clinicians pisiform contact. The force and vector applied will be the same.
  Other Names: Sham
  Arms: Sham Spinal Manipulation

SUMMARY:
The investigators propose a prospective randomized 2 arm parallel observer-blinded phase II clinical study comparing a distinct method of upper cervical chiropractic manipulation to a sham technique in 50 individuals with stage I hypertension (systolic blood pressure (SBP): 140-159 mm Hg; diastolic blood pressure (DBP):90-99 mm Hg).

DETAILED DESCRIPTION:
More than 50 million Americans suffer from hypertension, a disease with far-reaching public health impact causing or contributing to 7.1 million deaths yearly at an estimated annual incremental direct cost of $54 billion per year. Common treatments include antihypertensive medications and lifestyle modifications. While these treatments have been shown to be effective, only about 30% of hypertensive patients achieve blood pressure goals. Based on a recently published study (Bakris et al, 2007), one unique non-pharmaceutical approach may be a non-rotary type of upper cervical spinal manipulation to align the first cervical vertebra (atlas) performed by a doctor of chiropractic. We propose to conduct a similar study with a more commonly known chiropractic technique called Toggle Recoil. We propose a prospective randomized 2 arm parallel observer-blinded phase II clinical study comparing a distinct method of upper cervical chiropractic manipulation to a sham technique in 50 (25 in each group) individuals with Stage I hypertension (systolic blood pressure (SBP); 140-159 mm Hg or diastolic blood pressure (DBP):90-99 mm Hg). Patients will be seen by doctors of chiropractic twice each week for 6 weeks and outcomes will be collected at baseline, 3 weeks, and 6 weeks after enrollment. The primary outcome measure will be change in SBP and the primary endpoint will be at the week 6 assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 and < 75
* Documented Stage I Hypertension

Exclusion Criteria:

* Cardiovascular disorders (Angina pectoris, symptom of CHD; Hemodynamically significant valvular heart disease; Second or Third degree heart block without pacemaker; Stroke, MI, CV surgery within the past 12 months; Claudication, Aortic Coarctation)
* Defibrillator
* Autoimmune Arthropathies
* Pregnancy
* Unwillingness to stop other forms of manual therapy during study
* Unwillingness to sign ICD or preliminary consent
* Intention to move from the area during the next 4 months
* Unwillingness to participate in any of the treatment groups
* Avg SBP<140 or >159mm Hg (AND) Avg DBP<90 or >99mm Hg
* Any single SBP > 160mm Hg or DBP> 100
* BMI > 40
* Prescription medications with increased risk for CVA
* Current use of anti-coagulant medication/blood thinners
* Active drug or alcohol addiction or abstinent < 1 year
* Psychiatric diagnosis that would limit patient compliance
* Serious concomitant medical illness
* Contraindication(s) to treatment
* Electrolyte abnormalities seen on lab test
* Renal Failure w/ creatinine >2.5mg/dL
* Abnormal Liver function tests
* Anemia with hematocrit < 30%
* Glucose in Urine
* Serum potassium <3.4 @ baseline
* S/S Renal artery stenosis
* Quebec Task Force Classification 4-9
* Self-reported Arnold Chiari malformation
* Spinal or paraspinal tumors
* Dx with disorder that exhibit spinal joint hypermobility (Marfan Syndrome, Ehlers-Danlos Syndrome, Osteogenesis imperfecta)
* Unstable endocrine disorders
* Osteoporosis

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Goertz, DC, PhD, Principal Investigator — Palmer College of Chiropractic
Locations (1):
- Palmer College of Chirpractic, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Feasibility/pilot study

REFERENCES:
- [Background] Mansholt BA, Vining RD, Long CR, Goertz CM. Inter-examiner reliability of the interpretation of paraspinal thermographic pattern analysis. J Can Chiropr Assoc. 2015 Jun;59(2):157-64. PMID 26136608
- [Background] Hart JF. Effect of Spinal Manipulation of Upper Cervical Vertebrae on Blood Pressure: Results of a Pilot Sham-Controlled Trial. J Manipulative Physiol Ther. 2016 Oct;39(8):603. doi: 10.1016/j.jmpt.2016.08.008. Epub 2016 Oct 13. No abstract available. PMID 27745887
- [Background] Goertz CM, Salsbury SA, Vining RD. Response to Letter to the Editor on "Effect of Spinal Manipulation of Upper Cervical Vertebrae on Blood Pressure: Results of a Pilot Sham-Controlled Trial". J Manipulative Physiol Ther. 2016 Oct;39(8):603-604. doi: 10.1016/j.jmpt.2016.09.004. Epub 2016 Oct 11. No abstract available. PMID 27742418
- [Result] Goertz CM, Salsbury SA, Vining RD, Long CR, Pohlman KA, Weeks WB, Lamas GA. Effect of Spinal Manipulation of Upper Cervical Vertebrae on Blood Pressure: Results of a Pilot Sham-Controlled Trial. J Manipulative Physiol Ther. 2016 Jun;39(5):369-380. doi: 10.1016/j.jmpt.2016.04.002. Epub 2016 May 9. PMID 27157678
- See also: Inter-examiner reliability of the interpretation of paraspinal thermographic pattern analysis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4486995/

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Manipulation High Velocity: This non-rotary upper cervical procedure uses an impulse thrust with a controlled depth (high velocity). The participant's head is supported by a specially designed cushion and the doctor usually approaches the participant from in front of the head to contact soft tissue over the atlas transverse process, posterior to the lateral mass or occasionally on the C2 lamina or spinous process, with the pisiform process of one hand. The thrust is delivered by a contraction of the triceps muscles of both arms, which straightens the arms and applies the thrust to the participant.
  Spinal Manipulation is the application of a load (force or displacement) to specific body tissues (usually vertebral joints) with therapeutic intent. The mechanical characteristics of SM can vary in terms of its duration and amplitude, as well as its anatomical location, choice of levers, direction of force application, and the vehicle used to apply the force (manually or mechanically assisted).
Period: Overall Study
Arm/Group | Spinal Manipulation High Velocity | Sham Spinal Manipulation
Started | 24 | 27
Completed | 24 | 26
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spinal Manipulation High Velocity | Sham Spinal Manipulation | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (8.5) | 54.9 (12.1) | 56.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 15 | 15 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 20 | 42
  Black | 2 | 5 | 7
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Unadjusted and Adjusted Changes From Baseline in Systolic and Diastolic Blood Pressure at Weeks 1, 3, 6
Description: To estimate the effect size and variability of change in systolic (SBP) and/or diastolic blood pressure (DBP) over a six week treatment period to use in planning a full-scale randomized controlled trial and to assess the believability of the placebo manipulation.
  The table shows the unadjusted and adjusted mean change in SBP and DBP from baseline to after Treatment 1 (Tx 1), 3 (Wk 3), and 6 (Wk 6) Weeks.
  Adjusted values were adjusted for age, sex, BMI, and respective baseline blood pressure.
  Wk 3 and Wk 6 DBP were also adjusted for stage of blood pressure (prehypertension or Stage 1 hypertension).
Time Frame: Baseline after 1, 3, and 6 Weeks of treatment
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Spinal Manipulation High Velocity | Sham Spinal Manipulation
Number analyzed (Participants) | 24 | 27
mmHg
  Tx 1 - SBP (Unadjusted) | -1.2 [-4.8 to 2.5] | -5.3 [-8.7 to -1.8]
  Tx 1 - DBP (Unadjusted) | 0.8 [-1.3 to 2.9] | -1.7 [-3.7 to 0.3]
  Wk 3 - SBP (Unadjusted) | -3.6 [-7.8 to 0.7] | -3.3 [-7.4 to 0.8]
  Wk 3 - DBP (Unadjusted) | -2.4 [-5.2 to 0.3] | -2.2 [-4.8 to 0.4]
  Wk 6 - SBP (Unadjusted) | -0.1 [-4.0 to 3.8] | -3.6 [-7.3 to 0.2]
  Wk 6 - DBP (Unadjusted) | 0.3 [-2.2 to 2.9] | -1.2 [-3.6 to 1.3]
  Tx 1 - SBP (Adjusted) | -0.9 [-4.5 to 2.8] | -5.5 [-9.0 to -2.1]
  Tx 1 - DBP (Adjusted) | 1.4 [-0.7 to 3.4] | -2.2 [-4.2 to -0.3]
  Wk 3 - SBP (Adjusted) | -3.0 [-7.2 to 1.3] | -3.9 [-8.0 to 0.2]
  Wk 3 - DBP (Adjusted) | -1.8 [-4.5 to 0.9] | -2.8 [-5.4 to -0.2]
  Wk 6 - SBP (Adjusted) | 0.6 [-3.1 to 4.3] | -4.2 [-7.8 to -0.6]
  Wk 6 - DBP (Adjusted) | 0.7 [-1.7 to 3.2] | -1.6 [-3.9 to 0.8]
Statistical Analysis 1: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Tx 1 - SBP (Unadjusted); Test type: Other; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [-0.9 to 9.2]
Statistical Analysis 2: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Tx 1 - DBP (Unadjusted); Test type: Other; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-0.4 to 5.3]
Statistical Analysis 3: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Wk 3 - SBP (Unadjusted); Test type: Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-6.2 to 5.6]
Statistical Analysis 4: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Wk 3 - DBP (Unadjusted); Test type: Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-4.0 to 3.5]
Statistical Analysis 5: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Wk 6 - SBP (Unadjusted); Test type: Other; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-1.9 to 8.9]
Statistical Analysis 6: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Wk 6 - DBP (Unadjusted); Test type: Other; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-2.1 to 5.0]
Statistical Analysis 7: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Tx 1 - SBP (Adjusted); Test type: Other; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [-0.4 to 9.8]
Statistical Analysis 8: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Tx 1 - DBP (Adjusted); Test type: Other; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [0.6 to 6.5]
Statistical Analysis 9: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Wk 3 - SBP (Adjusted); Test type: Other; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-5.0 to 6.9]
Statistical Analysis 10: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Wk 3 - DBP (Adjusted); Test type: Other; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-2.8 to 4.9]
Statistical Analysis 11: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Wk 6 - SBP (Adjusted); Test type: Other; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-0.4 to 10.0]
Statistical Analysis 12: Comparison: Spinal Manipulation High Velocity vs Sham Spinal Manipulation; Wk 6 - DBP (Adjusted); Test type: Other; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-1.2 to 5.8]

2. Other Pre Specified Outcome: Number of Participants Who Were Recruited, Consented, Enrolled/Randomized, and Retained for the Duration of the Study
Description: To assess the feasibility of conducting a full-scale randomized controlled trial to evaluate the efficacy of Toggle Recoil chiropractic manipulation for patients with stage I hypertension. Feasibility measured by: patient recruitment, enrollment, and retention, and duration of study from launch date to final outcomes.
Time Frame: 19 months
Population: In this study, participants are not allocated to a treatment arm until they have met all eligibility criteria through the Final Case Review. Because of this it is not possible to report feasibility outcomes by treatment arm.
Measure: Number; unit: # participants
Groups:
- Feasibility Outcomes: Participants recruited, consented, enrolled, and retained, & duration of study from launch date to final outcomes.
Arm/Group | Feasibility Outcomes
Number analyzed (Participants) | 681
# participants
  # Participants screened via phone interview | 681
  # Participants consented at Baseline Visit 1 | 372
  # Participants eligible for final case review | 63
  # Participants Enrolled/Randomized | 51
  # Participants completed follow-up | 50

3. Other Pre Specified Outcome: Study Duration From Launch Date to Final Outcomes
Description: To assess the feasibility of conducting a full-scale randomized controlled trial to evaluate the efficacy of Toggle Recoil chiropractic manipulation for patients with stage I hypertension. Feasibility measured by and duration of study from launch date to final outcomes.
Time Frame: 19 months
Population: 51 participants were enrolled; however, the table below shows the number enrolled and consented before the 51 were enrolled. The final row of data shows, 19, signifying the study duration in MONTHS (October 2010 - April 2012).
Measure: Number; unit: months
Arm/Group | Feasibility Outcomes
Number analyzed (Participants) | 681
months | 19

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Any untoward medical occurrence that may present itself during the conduct of the study which may or may not have a causal relationship with the study procedures.
  *The total number of AEs may exceed the total # of people affected because some people experienced multiple AEs.
Groups:
- Spinal Manipulation High Velocity*: This non-rotary upper cervical procedure uses an impulse thrust with a controlled depth (high velocity). The participant's head is supported by a specially designed cushion and the doctor usually approaches the participant from in front of the head to contact soft tissue over the atlas transverse process, posterior to the lateral mass or occasionally on the C2 lamina or spinous process, with the pisiform process of one hand. The thrust is delivered by a contraction of the triceps muscles of both arms, which straightens the arms and applies the thrust to the participant.
  Spinal Manipulation is the application of a load (force or displacement) to specific body tissues (usually vertebral joints) with therapeutic intent. The mechanical characteristics of SM can vary in terms of its duration and amplitude, as well as its anatomical location, choice of levers, direction of force application, and the vehicle used to apply the force (manually or mechanically assisted).
- Sham Spinal Manipulation*: The sham assessment procedures will be similar to the active group. It has been developed and validated by Vernon et al.
  Sham Spinal Manipulation: The sham assessment procedures will be the same as those in the high velocity treatment group. The sham intervention is identical to this treatment protocol except for the placement of the treating clinicians pisiform contact. The force and vector applied will be the same.
Arm/Group | Spinal Manipulation High Velocity* | Sham Spinal Manipulation*
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 6/24 | 5/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spinal Manipulation High Velocity* (N=24) | Sham Spinal Manipulation* (N=27)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Musculoskeletal and connective tissue disorders) | 2 | 0
Migraine (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache and tenderness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck and back pain and fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Radiating symptoms (General disorders) | 0 | 2
Dizziness/imbalance/vertigo (General disorders) | 0 | 1
Hypertension (General disorders) | 0 | 1
Hypotension (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes